CLINICAL TRIAL: NCT00092287
Title: A Phase III, Prospective, Multicenter, Randomized, Open, Parallel Group Comparison of Lanreotide Autogel® (90 and 120 mg) Administered by Deep Subcutaneous Injection Every Four Weeks, With Sandostatin LAR Depot (20 and 30 mg) Administered by Intramuscular Injection, Every Four Weeks for Six Months, in the Treatment of Clinical Symptoms Associated With Carcinoid Syndrome
Brief Title: Comparison of Lanreotide Autogel® and Sandostatin LAR Depot in the Treatment of Clinical Symptoms Associated With Carcinoid Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-47-52030-722; 2004-001091-40 (EudraCT Number)
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Malignant Carcinoid Syndrome
Keywords: Carcinoid Syndrome; Neuroendocrine Tumuors
MeSH Terms: conditions — Malignant Carcinoid Syndrome; Serotonin Syndrome | interventions — Receptor-Like Protein Tyrosine Phosphatases, Class 2

INTERVENTIONS:
Drug: lanreotide Autogel (somatostatin analogue)
Drug: Sandostatin long acting release (LAR) Depot (somatostatin analogue)

SUMMARY:
The aim of this study is to compare the efficacy and safety of lanreotide Autogel and Sandostatin LAR Depot, to see whether these two 28-day prolonged release formulations produce a similar clinical response in patients with carcinoid syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a neuroendocrine tumor of the carcinoid type.
* Documented evidence of carcinoid syndrome (flushing and/or diarrhea) attributable to a primary tumor of the lung, stomach or mid-gut.
* Previous positive Octreoscan.
* World Health Organization (WHO) performance score lower than 2.

At the baseline visit patients MUST satisfy the following criteria before they are randomized to receive study treatment:

* Stool and/or flushing frequency of greater than or equal to 3 episodes/day (average over a minimum five consecutive days).
* Patients who have previously been treated with somatostatin analogues must have discontinued treatment for a sufficient period of time (a washout period of at least 7 days for immediate release formulations and up to 2 months for prolonged release formulations is usually required). Compared with their "controlled" state on treatment, these patients must show a clinically significant deterioration (at least two episodes) of either symptom. For example, a patient considered to be controlled on their previous treatment with an estimated stool frequency of two episodes per day, must achieve a stool frequency of at least four episodes per day (average over a minimum five consecutive days).
* WHO performance score lower than 2.

Exclusion Criteria:

* VIPoma or other non-carcinoid tumor.
* Treatment with interferon, chemotherapy or radiotherapy given within 30 days prior to inclusion, or planned during the study.
* Radionuclide treatment within three months prior to inclusion, or planned during the study.
* Presence of other active malignant pathology (except basal cellular carcinoma of the skin and/or in situ carcinoma of the cervix/uterus).
* Surgical procedure or embolization procedure (with or without cytotoxic agents) of the tumor within three months prior to inclusion, or planned during the study.
* Life expectancy of less than 6 months.
* Any investigational drug given within 30 days prior to inclusion or expected to be given during the study.
* No access to a telephone for completion of the daily telephone diary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-07; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Target symptom frequency (flushing or stool frequency).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Larry Kvols, MD, Tampa, Florida, United States